CLINICAL TRIAL: NCT03690570
Title: Long Term Follow up of Patients Under 5 Years of Age With High Grade Glioma Diagnosed in France Between 1990 and 2015
Acronym: GlioUnder5
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6964
Record Dates: First submitted 2018-06-28; First posted 2018-10-01 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-06

CONDITIONS: Glioma
Keywords: Glioma; Children; Chemotherapy; treatment toxicitT; Survival
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High grade glioma is a rare disorder affecting children at all ages with a high mortality rate. Overall survival is estimated at 40%, depending on the type of treatment administered. Major late sequelaes are experienced with the irradiation in this population under 5 years. Therefore, the current recommendations by The French Society for Childhood Cancers are based on a treatment including surgery followed by chemotherapy and avoiding radiotherapy as long as patients present no sign of treatment failure. The results published in 2006, underlying the fact that some patients treated exclusively with surgical resection and chemotherapy can achieve long term survival, are showing evidence of an acceptable long-term strategy. Few studies concerning evaluation of treatment toxicity and long term outcomes are available. Therefore, it is important to collect retrospective data concerning those small patients with high grade glioma in order to understand the reasons of treatment success or failure and treatment toxicities. This retrospective study will evaluate long term survivals comparatively to clinical, radiological and histological features at diagnosis and the treatment toxicities including neurological, endocrine and hearing impairment to go further and propose new potential guidelines and chemotherapy schedules

ELIGIBILITY:
Inclusion Criteria:

* Children under 5 years old
* High grade glioma (WHO status III or IV)
* No previous treatment with chemotherapy or radiotherapy
* No contraindication to chemotherapy
* Consent of legal representative for participation in the study

Exclusion Criteria:

* Low grade glioma
* Any other histological pattern
* Parent's denial to access data concerning their child in the frame of medical research

Ages: 1 Day to 5 Years | Sex: All
Age Groups: Child
Study Population: Children under 5 years old with high grade glioma (WHO status III or IV)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-05-09 (Estimated); Study Completion 2019-05-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of patient survival associated with relapse rate after surgery | 10 years
Assessment of patient survival associated with relapse rate after chemotherapy | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Natacha ENTZ-WERLE, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Pédiatrie 3, Strasbourg, France